CLINICAL TRIAL: NCT00773448
Title: Screening for Occult Malignancy in Patients With Idiopathic Venous Thromboembolism: an Open Randomized Controlled Trial Using a Comprehensive Abdomen/Pelvis Computed Tomography
Brief Title: Screening for Occult Malignancy in Patients With Idiopathic Venous Thromboembolism
Acronym: SOME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Marc Carrier, MD, MD MSc FRCPC, Scientist., Ottawa Hospital Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2004723-01H
Record Dates: First submitted 2008-10-14; First posted 2008-10-16 (Estimated); Last update posted 2015-07-07 (Estimated); Status verified 2015-07

CONDITIONS: Venous Thromboembolism; Deep Vein Thrombosis; Pulmonary Embolism
Keywords: Cancer; Screening
MeSH Terms: conditions — Venous Thromboembolism; Venous Thrombosis; Pulmonary Embolism; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Limited Malignancy Screening (Active Comparator)
  Interventions: Other: Limited Malignancy Screening
- Extensive Malignancy Screening (Experimental): Limited screen as described above in combination with comprehensive computed tomography of the abdomen/pelvis
  Interventions: Device: Comprehensive computed tomography of the abdomen/pelvis

INTERVENTIONS:
Device: Comprehensive computed tomography of the abdomen/pelvis — Virtual colonoscopy and gastroscopy, a biphasic enhanced CT for hepatoma and renal cell carcinoma, parenchymal pancreatogram with minimum intensity projection (MinIP) reformation for pancreatic carcinoma, and finally uniphasic enhanced CT of distended bladder for bladder and ovarian carcinomas.
  Arms: Extensive Malignancy Screening
Other: Limited Malignancy Screening — 1) A complete medical history and physical examination; 2) complete blood count; 3) liver function tests (AST, ALT, ALP, bilirubin, LDH); 4) renal function test (creatinine); 5) chest X-ray (if not performed in the past year)
  In women, a pap smear/pelvic examination (if > 18 and < 70 years old and not performed during the past year),a mammogram (> 50 years old) will be performed if not conducted in last year. Similarly for men, prostate examination +/- PSA testing (>40 years old) will be performed if not conducted in the past year.
  Arms: Limited Malignancy Screening

SUMMARY:
Blood clots in leg veins (deep vein thrombosis) or lung arteries (pulmonary embolism) that happen for no reason (i.e. unexplained) are both called "unprovoked venous thromboembolism" (VTE). These unexplained blood clots can be the first symptom of cancer. Up to 10% of patients with unexplained blood clots will be diagnosed with cancer within one year of their blood clot diagnosis.

These cancers can be found anywhere in the body although the relationship appears stronger with the pancreas, ovary and liver. Cancer testing in patients with blood clots is controversial. There is presently a wide variety of expert opinions and practices. Previous studies showed that a limited cancer screen including a medical history, physical examination, basic blood work and chest X-ray, will find about 90% of cancers. More recent and better designed studies showed that the limited cancer screen misses many cancers and needs to be improved. More extensive cancer testing may find more cancers but is potentially uncomfortable for patients, costs a lot of money and involves a lot of people.

The "comprehensive computed tomography" is less uncomfortable, inexpensive, radiological test made to find many cancers at once. Thus, the scientific question to be asked is: Does a "comprehensive computed tomography" miss less cancers than a limited cancer screen in patients with blood clots?

The main goal of this study is to find out if a "comprehensive computed tomography" misses less cancers than a limited cancer screen in patients with unexplained blood clots.

The second goal of the study is 1) to find out if a "comprehensive computed tomography" finds more "curable" cancers than the limited cancer screen; 2) to find out if the patients diagnosed with cancer are still alive and cancer-free after one year (i.e. the patients with curable cancer were treated and are doing well); 3) to prove that a negative "comprehensive computed tomography" means that the patient will not have cancer and; 4) to find out if a "comprehensive computed tomography" is well tolerated and safe for patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a new diagnosis of unprovoked proximal deep vein thrombosis (DVT) or pulmonary embolism (PE) will be eligible to participate into the study:

  * Unprovoked VTE is defined as the absence of any of the following predisposing factors:

    1. known active cancer;
    2. recent (less than 3 months) paralysis, paresis or plaster immobilization of the lower extremities;
    3. recently bedridden for period of 3 or more days, or major surgery, within the previous 12 weeks requiring general or regional anaesthesia;
    4. previous unprovoked VTE;
    5. known thrombophilia (hereditary or acquired)
  * Proximal DVT is defined as a non-compressibility of any vein segment from the common femoral vein to the trifurcation of the popliteal vein or a persistent intra-luminal filling defect of the iliac, common femoral, superficial femoral or popliteal veins on contrast venography.
  * Pulmonary embolism is defined as:

    1. patients with a high/intermediate pre-test probability (Wells' model > 4) + high probability V/Q scan;
    2. positive pulmonary angiogram; or
    3. spiral CT demonstrating intraluminal filling defect in a vessel larger than a segmental artery

Exclusion Criteria:

Patients will be excluded from the study if they have any of the following criteria:

* Age < 18 years-old;
* Refusal or inability to provide informed consent;
* Greater than 21 days post diagnosis of idiopathic VTE
* Index VTE event of UEDVT or unusual site DVT
* Diagnosis of SSPE in the absence of above or below knee DVT
* Allergy to contrast media;
* Creatinine clearance < 60 ml/min;
* Claustrophobia or agoraphobia;
* Weight > 130 kg;
* Diagnosis of ulcerative colitis; and
* Diagnosis of glaucoma
* Current pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 862 (Actual)
Dates: Start 2008-09; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Previously undiagnosed malignancy "missed" by malignancy screening defined as biopsy proven tissue diagnosis of malignancy diagnosed from the time of malignancy screening completion to the end of the 1 year follow-up period. | 1 year

SECONDARY OUTCOMES:
Overall mortality | 1 year
Recurrent VTE | 1 year
Early malignancy: T1-2N0M0 as per the World Health Organization TNM classification system | 1 year
QALYs gained | 1 year
Incremental cost-effectiveness ratio | 1 year
Adverse events with cCT | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Marc Carrier, MD MSc FRCPC, Principal Investigator — The Ottawa Hospital Research Institute
Locations (9):
- Canada (9):
  - St. Boniface Hospital, Winnipeg, Manitoba
  - Capital Health Centre for Research, Halifax, Nova Scotia
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - London Health Sciences Center, London, Ontario
  - Ottawa Hospital, Ottawa, Ontario
  - Montreal General Hospital, Montreal, Quebec
  - Sacre-Coeur Hospital, Montreal, Quebec
  - Sir Mortimer B. Davis Jewish General Hospital, Montreal, Quebec
  - St. Mary's Hospital Center, Montreal, Quebec

REFERENCES:
- [Background] Carrier M, Le Gal G, Wells PS, Fergusson D, Ramsay T, Rodger MA. Systematic review: the Trousseau syndrome revisited: should we screen extensively for cancer in patients with venous thromboembolism? Ann Intern Med. 2008 Sep 2;149(5):323-33. doi: 10.7326/0003-4819-149-5-200809020-00007. PMID 18765702
- [Result] Carrier M, Lazo-Langner A, Shivakumar S, Tagalakis V, Zarychanski R, Solymoss S, Routhier N, Douketis J, Danovitch K, Lee AY, Le Gal G, Wells PS, Corsi DJ, Ramsay T, Coyle D, Chagnon I, Kassam Z, Tao H, Rodger MA; SOME Investigators. Screening for Occult Cancer in Unprovoked Venous Thromboembolism. N Engl J Med. 2015 Aug 20;373(8):697-704. doi: 10.1056/NEJMoa1506623. Epub 2015 Jun 22. PMID 26095467
- [Derived] Robertson L, Broderick C, Yeoh SE, Stansby G. Effect of testing for cancer on cancer- or venous thromboembolism (VTE)-related mortality and morbidity in people with unprovoked VTE. Cochrane Database Syst Rev. 2021 Oct 1;10(10):CD010837. doi: 10.1002/14651858.CD010837.pub5. PMID 34597414
- [Derived] Ihaddadene R, Corsi DJ, Lazo-Langner A, Shivakumar S, Zarychanski R, Tagalakis V, Solymoss S, Routhier N, Douketis J, Le Gal G, Carrier M. Risk factors predictive of occult cancer detection in patients with unprovoked venous thromboembolism. Blood. 2016 Apr 21;127(16):2035-7. doi: 10.1182/blood-2015-11-682963. Epub 2016 Jan 27. PMID 26817957